CLINICAL TRIAL: NCT05402059
Title: prospectIve Non-interventional Study of Clinical Outcomes And Biomarkers in Patients With Stage 0-IV mElanoma in reaL clinicaL prActice
Brief Title: Clinical Outcomes and Biomarkers in Patients With Stage 0-IV Melanoma in Real Clinical Practice
Acronym: ISABELLA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MelanomaPRO, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: MELPRO-0921
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Melanoma; Melanoma (Skin); Melanoma, Uveal; Melanoma Stage IV; Melanoma Stage III; Melanoma, Stage II; Melanoma in Situ; Melanoma, Ocular
MeSH Terms: conditions — Melanoma; Uveal Melanoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin fixed paraffin embedded tumor tissue blocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort A: Study Cohort A will include patients with unresectable and/or metastatic melanoma, regardless of BRAF mutation in the tumor, who were started on any of the drug regimens in accordance with current clinical guidelines, except for patients assigned to the vemurafenib + cobimetinib + atezolizumab, which should be included in the A1 cohort. The initiation of therapy on the regimen that will be used at the time of signing the informed consent will be considered an index event.
  Interventions: Drug: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines
- Cohort A1: Study Cohort A1 will include patients with unresectable and/or metastatic melanoma and an activating BRAF mutation in the tumor who were treated with vemurafenib + cobimetinib + atezolizumab, either newly diagnosed or progressing during previous lines of therapy. Initiation of vemurafenib + cobimetinib + atezolizumab would be considered an index event.
  Interventions: Drug: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines
- Cohort B: Study Cohort B will include patients with stage III equivalent skin melanoma (i.e., regional lymph node involvement), regardless of tumor BRAF mutation, who have undergone surgery (lymphadenectomy, SLNB, or metastasectomy) and/or initiated or planned treatment according to any of the drug therapy regimens or only dynamic observation, in accordance with current clinical guidelines. Surgery for stage III melanoma will be considered an index event.
  Interventions: Drug: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines
- Cohort C: Study cohort C will include patients with stage 0-II equivalent skin melanoma (i.e., no regional lymph node involvement), regardless of BRAF mutation in the tumor, who have undergone surgery (excision of the primary tumor +/- SLNB) and/ or initiated or planned treatment for any of the drug regimens or only dynamic observation, in accordance with current clinical guidelines. Surgical treatment (operation) for stage 0-II melanoma will be considered an index event.
  Interventions: Drug: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines
- Cohort D: Study cohort D will include patients with stage 0-IV non-cutaneous melanoma, regardless of the BRAF mutation in the tumor, who underwent morphological verification of the diagnosis, surgery (any volume) and / or treatment initiated or planned for any of the drug therapy regimens or only dynamic observation, in accordance with current clinical guidelines. Initiation of therapy according to the regimen that will be used at the time of signing of informed consent or surgical treatment will be considered an index event.
  Interventions: Drug: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines

INTERVENTIONS:
Drug: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — Any kind of treatment or observation (no treatment) initiated or planned in accordance with current clinical practice

SUMMARY:
Prospective non-interventional study of clinical outcomes and biomarkers in patients with stage 0-IV skin melanoma in real clinical practice

DETAILED DESCRIPTION:
Most oncology experts now recognize that the most effective and safest treatment options should be considered for first-line therapy. Since the planned use of drugs, including dosing, treatment interruption and early discontinuation of treatment, in clinical practice may differ from the procedures used in clinical trials, post-marketing "real world" data are important to quantify the feasibility, acceptability, and practical considerations for prescribing targeted and immunotherapy. Therefore, for the clinical and scientific communities, it is of great interest to evaluate the choice of the patient and the method of treatment used in the daily practice of oncological centers in Russia. Moreover, the available data imply an association between PDl-1 expression and other biomarkers in tumors and the efficacy of drug therapy. The purpose of this study is to evaluate clinical outcomes in patients with stage 0-IV skin melanoma in real clinical practice in the context of different levels of PDl-1 expression in the tumor and other potential biomarkers. In addition, it is of interest to gain insight into the real-world data on the quality of life of melanoma patients treated for metastatic disease. It is well known, that the prognosis of patients with stage 0-IV melanoma is too heterogeneous, therefore, in this study, distinguish several cohorts will be organised.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria (all cohorts):

* male or female patients 18 years of age or older;
* ECOG status <=3;
* the current treatment regimen (index date) was started no earlier than 12 weeks (84 days) prior to obtaining written informed consent to participate in this study;
* patients who are willing and able to participate in the study;
* informed consent to participate in the study was obtained.

Inclusion criteria for cohort A:

-Confirmed by histopathology cutaneous melanoma stage IV metastatic cutaneous melanoma (or IIIC/D unresectable stage or cutaneous melanoma metastases without a primary lesion or equivalent) with or without a BRAF mutation for which the attending physician has decided to initiate any systemic or local treatment before inclusion in the study;

Inclusion criteria for cohort A1:

* Confirmed by histopathology stage IV (or unresectable stage IIIC/D or non-resectable cutaneous melanoma metastases or equivalents) with a confirmed BRAF mutation for which the treating physician has decided to initiate treatment with vemurafenib + cobimetinib + atezolizumab before inclusion in study;
* treatment with vemurafenib + cobimetinib + atezolizumab was started no earlier than 12 weeks (84 days) prior to obtaining written informed consent to participate in this study;

Inclusion criteria for cohort B:

- Confirmed by histopathology melanoma of the skin with regional lymph node involvement, transit or satellite metastases (equivalent to IIIA, B, C/D resectable stage) with or without a BRAF mutation, for which the attending physician decided to start any systemic or local treatment before enrollment in the study ;

Inclusion criteria for cohort C:

* Confirmed by histopathology melanoma of the skin melanoma of the skin without involvement of regional lymph nodes, without clinically or morphologically determined transit or satellite metastases (equivalent to 0-IIC resectable stage) with or without a BRAF mutation, about which the attending physician has decided to start any systemic or local treatment before inclusion in the study;
* Skin melanoma thicker than 0.8 mm Breslow was staged with a sentinel lymph node biopsy procedure;

Inclusion criteria for cohort D:

• Confirmed by histopathology or cytology non-cutaneous melanoma of any stage (including but not limited to patients with melanoma of the mucous membranes of the upper respiratory and digestive tract, anal canal, female and male genital organs, choroid), for which the attending physician has decided to start any systemic or topical treatment before inclusion in the study;

Exclusion Criteria:

* Patients with a life expectancy of less than 1 month at the time of diagnosis of melanoma, according to the investigator.
* Patients enrolled in any interventional clinical trial involving the use of experimental drugs or drugs available over the counter at the time of enrollment in the study. (Patients enrolled in another investigator-initiated study or non-interventional study may be included in this study if it does not involve changes to their standard of care.)
* Patients with no histologically confirmed diagnosis of melanoma and who are receiving active treatment for cancers other than melanoma at the time of enrollment. Patients with multiple primary synchronous or metachronous tumors, at least one of which is melanoma, may be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study will be conducted in investigation sites specialized in treatment of solid neoplasm or, more narrowed, melanoma. Patient may be enrolled either by surgical or medical oncologist if relevant indormation is available and there is no obvious risk for loss of contact with patient. Study population will be formed of the patients from cancer treatment facilities and the representativeness of sample may vary depending on participating sites.
Sampling Method: Probability Sample
Enrollment: 1570 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
12-month relapse-free survival | 12 months
  The primary efficacy endpoint of the study is 12-month relapse-free survival, defined as the time from index date to the date of first documented relapse or death from any cause (for stage 0-III asymptomatic patients with or without adjuvant therapy, cohorts B and C).
12-month progression free survival | 12 months
  The second primary efficacy endpoint is the 12-month PFS, defined as the time from the index date to the date of the first documented investigator-determined progression or death from any cause. If the patient has not experienced an event, PFS will be censored at the date of the last tumor assessment (for patients with IIIC/D unresectable or metastatic melanoma, cohorts A, A1, D).

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin Russian Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Samoylenko IV, Kolontareva YM, Kogay EV, Zhukova NV, Utyashev IA, Ivannikov ME, Menshikov KV, Zinkevich MV, Orlova KV, Vakhabova YV, Volkonsky MV, Beliaeva NA, Butkov II, Karabina EV, Moskovkina TL, Moshkova KA, Plishkina OV, Sychev VD, Cheplukhova OS, Chernova VV, Yurchenkov AN, Babina KG, Savelov NA, Demidov LV. Triple combination of vemurafenib, cobimetinib, and atezolizumab in real clinical practice in the Russian Federation: results of the A1 cohort of the ISABELLA study. Front Oncol. 2024 Oct 14;14:1395378. doi: 10.3389/fonc.2024.1395378. eCollection 2024. PMID 39469641